CLINICAL TRIAL: NCT04079738
Title: Phase I/II Study Augmenting TAK-659 Action in Relapsed/Refractory AML by Addition of the Proteasome Inhibitor Ixazomib: Big Ten Cancer Research Consortium BTCRC-HEM17-092
Brief Title: Study Augmenting TAK-659 Action in Relapsed/Refractory AML by Addition Ofthe Proteasome Inhibitor Ixazomib
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funder requested termination due to halting internal development of TAK-659
Sponsor: H Scott Boswell (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, H Scott Boswell, Professor, Department of Medicine, Division of Hematology/Oncology, IU School of Medicine, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-HEM17-092
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: AML; AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — TAK-659; ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I:TAK-659 + Ixazomib (Experimental): Phase I: TAK-659 (Days 1-15) + Ixazomib dose escalation (Days 1, 8, 15)
  Interventions: Drug: TAK-659; Drug: Ixazomib
- Phase II:TAK-659 + Ixazomib (Experimental): Phase II: TAK-659 at MTD (Days 1-15) + Ixazomib at MTD (Days 1, 8, 15)
  Interventions: Drug: TAK-659; Drug: Ixazomib

INTERVENTIONS:
Drug: TAK-659 — TAK-659
Drug: Ixazomib — Ixazomib

SUMMARY:
This is a Phase I/II study augmenting TAK-659 action in relapsed/refractory AML by addition of the proteasome inhibitor Ixazomib. Phase I of the study will determine the safety, tolerability, and maximum tolerated dose (MTD) of the combination of TAK-659 and Ixazomib. During the phase I, dose escalation will be conducted according to a standard 3+3 dose escalation schema, and up to 18 response-evaluable patients will be enrolled. Phase II of the study will evaluate the efficacy of the combination by measuring the overall response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Male or female patients 18 years or older at the time of consent.
* Patients must have a diagnosis of primary or secondary AML with relapsed or refractory disease (WHO update 2016, [34]) other than acute promyelocytic leukemia, or complex karyotype or monosomy 7 (or containing monosomy 7) for whom no standard therapies are anticipated to result in a durable remission according to the clinical judgment of the treating physician, or in a patient who refuses standard therapies.
* Must have submitted for Next Generation Sequencing (NGS) testing by: 1) (preferred) having submitted a tumor sample for commercial myeloid NGS from Foundation One, Mayo, Tempus, Quest, ARUP or an institutional CLIA-certified laboratory and/or 2) obtaining a bone marrow aspirate during screening for submission to Foundation One, Mayo, Tempus, Quest, ARUP or an institutional CLIA-certified laboratory and ordered as standard of care. If bone marrow aspiration has failed, a peripheral blood sample with circulating blasts may be substituted. Screening reports on tumor cytogenetics and/or mutation assays (eg, FLT-3, and NGS) performed as part of the standard of care will be recorded in the study database or obtained at the time of screening if not previously available.
* Patient's disease must be characterized for the presence/absence of Flt3ITD/TKD mutation from an FDA-approved vendor (ex. LabPMM).
* In addition, patients for the phase 2 portion of the study must meet the following:

  * Patients, if relapsed/ refractory, must have exposure to no more than 2 prior chemotherapy regimens. Re-induction with the same regimen or stem cell transplant will not be considered a separate regimen.
  * Patients must not have prior exposure to any investigational Flt3 inhibitors (midostaurin or gilteritinib are allowed)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of greater than 3 months as determined by the treating physician.
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception at the same time, from the time of signing the informed consent through 180 days after the last dose of study drug, or
  * Agree to practice true abstinence, when is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
  * Agree not to donate eggs (ova) during the course of this study or 180 days after receiving their last dose of study drug.
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 180 days after the last dose of study drug, or
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception. Female and male condoms should not be used together.)
  * Agree not to donate sperm during the course of this study or within 180 days after receiving their last dose of study drug.
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* In the absence of rapid progressive disease, the interval from prior systemic anticancer treatment to time of TAK-659/Ixazomib administration should be at least 2 weeks for cytotoxic agents (other than hydroxyurea), or at least 5 half-lives for noncytotoxic agents, and patients have to have recovered from acute toxicities of these therapies. Patients who are on hydroxyurea may be included in the study and may continue on hydroxyurea for the first 21 days while participating in this study. NOTE: For patients with a white blood cell count >50,000/uL, hydroxyurea may be used to control the level of circulating leukemic blast cell counts prior to study entry, and, if needed, concomitantly while on TAK-659 treatment during the first 21 days of the study.
* Suitable venous access for the study-required blood sampling, and transfusion support.
* Demonstrate adequate organ function as defined in the protocol; all screening labs to be obtained within 28 days prior to registration.

Exclusion Criteria:

* Clinically active central nervous system leukemia.
* Female patients who are lactating and breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study)
* Female patients who have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
* Any serious medical or psychiatric illness, including drug or alcohol abuse, that could, in the investigator's opinion, potentially jeopardize the safety of the patient or interfere with the objectives of the study.
* Prior treatment with investigational agents ≤ 21 days or ≤ 5 half-lives (whichever is shorter) before the first dose of study treatment. A minimum of 10 days should elapse from prior investigational therapy to initiating protocol therapy.
* Persistent clinically significant toxicity from prior chemotherapy that is Grade 2 or higher by the NCI CTCAE (v5).
* Receipt of HSCT within 60 days of the first dose of TAK-659/Ixazomib; clinically significant graft-versus-host disease (GVHD) requiring ongoing immunosuppressive therapy post HSCT at the time of screening (use of topical steroids for ongoing skin GVHD is permitted).
* Active, systemic infection requiring intravenous (IV) antibiotic, antifungal, or antiviral therapy or other serious infection within 10 days before the first dose of study drug.
* Major surgery within 14 days before the first dose of study drug and have not recovered fully from any complications from surgery.
* Radiotherapy less than 2 weeks before the first dose of study treatment or have not recovered from acute toxic effects from radiotherapy.
* Known human immunodeficiency virus (HIV) positive.
* Known hepatitis B surface antigen positive, or known or suspected active hepatitis C infection (testing not required).
* Any of the following cardiovascular conditions:

  * Acute myocardial infarction within 6 months before starting study drug.
  * Current or history of New York Heart Association Class III or IV heart failure (see Study Procedures Manual [SPM]).
  * Evidence of current, uncontrolled cardiovascular conditions including cardiac arrhythmias, angina, pulmonary hypertension, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
  * Fridericia corrected QT interval (QTcF) >450 milliseconds (msec) (men) or >475 msec (women) on a 12-lead ECG during the Screening period.
  * Abnormalities on 12-lead ECG including, but not limited to, changes in rhythm and intervals that, in the opinion of the treating physician, are considered to be clinically significant.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance to study drugs, including difficulty swallowing tablets, diarrhea > Grade I despite supportive therapy.
* Use or consumption of any of the following medications, supplements, or foods/beverages that are inhibitors or inducers of P-gp or strong reversible inhibitors or inducers of CYP3A within the indicated timeframes below. Note that use or consumption of these substances is not permitted during the study.

  * Inhibitors of P-gp and/or strong reversible inhibitors of CYP3A within 5 times the inhibitor half-life (if a reasonable half-life estimate is known), or within 7 days (if a reasonable half-life estimate is unknown), before the first dose of study drug. In general, the use of these agents is not permitted during the study except in cases where an AE must be managed. See SPM for a nonexhaustive list of strong CYP3A reversible inhibitors and/ or Pgp inhibitors based on the FDA Draft DDI Guidance.
  * Strong CYP3A mechanism-based inhibitors or strong CYP3A inducers and/or P-gp inducers within 7 days, or within 5 times the inhibitor or inducer half-life (whichever is longer), before the first dose of study drug. However, if a patient has a strong indication for fungal prophylaxis, then the moderate CYP3A inhibitors fluconazole or isovuconazole (mold-active) is recommended for prophylaxis, and the TAK-659 dose should be reduced to 60mg, along with increased scrutiny for toxicity. Similarly, if the patient develops a fungal infection during a productive intervention with TAK-659/Ixazomib combination, isovuconazole (mold-active) should be used, along with increased scrutiny for toxicity. In general, the use of these agents is not recommended during the study except in cases where such an AE must be managed, and the intermittent schedule of TAK-659/Ixazomib combination will not prevent profound neutropenia. See SPM for a non-exhaustive list of strong CYP3A mechanism-based inhibitors or strong CYP3A inducers and/or P-gp inducers based on the FDA Draft DDI Guidance.
  * Grapefruit-containing food or beverages within 5 days before the first dose of study drug.
* Lack of suitable venous access for the study-required blood sampling.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient has Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H Scott Boswell, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Level 1: TAK-659 100mg + Ixazomid 2.3mg: Phase I,Level 1: TAK-659 100mg (Days 1-15) + Ixazomib 2.3mg dose escalation (Days 1, 8, 15)
  TAK-659: Subjects were given 100 mg of TAK-659 tablets once daily for fifteen days.
  Ixazomib: Subjects were given 2.3 mg of Ixazomib capsules once weekly on days 1, 8,15, respectively.
- Phase I, Level 2: TAK-659 100mg + Ixazomid 3mg: Phase I,Level 2: TAK-659 100mg (Days 1-15) + Ixazomib 3mg dose escalation (Days 1, 8, 15)
  TAK-659: Subjects were given 100 mg of TAK-659 tablets once daily for fifteen days.
  Ixazomib: Subjects were given 3 mg of Ixazomib capsules once weekly on days 1, 8,15, respectively.
- Phase I, Level 3: TAK-659 100mg + Ixazomid 4mg: Phase I, Level 3: TAK-659 100mg (Days 1-15) + Ixazomib 4mg dose escalation (Days 1, 8, 15)
  TAK-659: Subjects were given 100 mg of TAK-659 tablets once daily for fifteen days.
  Ixazomib: Subjects were given 4 mg of Ixazomib capsules once weekly on days 1, 8,15, respectively.
- Phase II:TAK-659 100mg+ Ixazomib MTD: Phase II: TAK-659 100 mg (Days 1-15) + Ixazomib at MTD (Days 1, 8, 15)
  TAK-659: Subjects were given 100 mg ofTAK-659 tablets once daily for fifteen days at MTD.
  Ixazomib: Subjects were given Ixazomib capsules once weekly at MTD on days 1, 8,15, respectively at MTD.
Period: Study Treatment
Arm/Group | Phase I, Level 1: TAK-659 100mg + Ixazomid 2.3mg | Phase I, Level 2: TAK-659 100mg + Ixazomid 3mg | Phase I, Level 3: TAK-659 100mg + Ixazomid 4mg | Phase II:TAK-659 100mg+ Ixazomib MTD
Started | 8 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — withdrawal before treatment | 1 | 0 | 0 | 0
Not completed — symptomatic deterioration | 2 | 0 | 0 | 0
Not completed — Disease Progression | 1 | 0 | 0 | 0
Not completed — withdrawal after treatment | 1 | 0 | 0 | 0
Period: Follow up
Arm/Group | Phase I, Level 1: TAK-659 100mg + Ixazomid 2.3mg | Phase I, Level 2: TAK-659 100mg + Ixazomid 3mg | Phase I, Level 3: TAK-659 100mg + Ixazomid 4mg | Phase II:TAK-659 100mg+ Ixazomib MTD
Started | 8 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Not completed — Death | 5 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There was one patient who had been eligible but never received treatment. The seven subjects who received active study treatment have been considered in this baseline analysis population.
  This study was terminated due to Funder's decision during Phase I portion of the study.
Arm/Group | Phase I, Level 1: TAK-659 100mg + Ixazomid 2.3mg
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 7
  Race: Unknown | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic | 7
  Ethnicity: Unknown | 0
ECOG PS at screening [Count of Participants; unit: Participants] — ECOG performance scores can be explained as follows:
  0: Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  Participants
    1 | 3
    0 | 4
Cigarette Usage [Count of Participants; unit: Participants]
  Never a smoker | 5
  Former smoker | 2
  Current smoker | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose(s) (RP2D)
Description: To determine the maximum tolerated dose (MTD) and recommended phase 2 dose(s) (RP2D) of the combination of TAK-659 and Ixazomib in patients with relapsed or refractory AML.
Time Frame: At the end of Cycle 2(each cycle is 28 days)
Measure: Number; unit: mg
Groups:
- Phase I: TAK-659 100mg + Ixazomid 2.3mg: TAK-659 100mg + Ixazomib 2.3mg
  TAK-659: Subjects were given 100 mg ofTAK-659 tablets once daily for fifteen days at MTD.
  Ixazomib: Subjects were given Ixazomib capsules 2.3 mg, on days 1,8,15
Arm/Group | Phase I: TAK-659 100mg + Ixazomid 2.3mg
Number analyzed (Participants) | 8
mg | NA — Maximum Tolerated Dose (MTD) was not determined due to the early termination of the trial by the funder. All subjects were treated with the first dose level.

2. Primary Outcome: Overall Response Rate for Phase II Subjects.
Description: To evaluate preliminary efficacy of TAK-659 plus Ixazomib in relapsed or refractory AML as measured by overall response rate (ORR).
  Overall response rate (ORR) defined as CR, CRp, CRi, and PR per Revised Recommendations of the International Working Group (IWG) for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia.
Time Frame: Overall Response rate is assessed at the end of 4 cycles ; 4 months.
Population: This study was terminated due to Funder's decision at Phase I.
Arm/Group | Phase II:TAK-659 100mg+ Ixazomib MTD
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DOR) for Phase II Subjects
Description: DOR defined as the time from the date of first documentation of a response to the date of first documented progressive disease
Time Frame: Up to two years after the date of the first documented response.
Population: The study was terminated at phase I due to Funder's decision.
Arm/Group | Phase II:TAK-659 100mg+ Ixazomib MTD
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression (TTP) for Phase II Subjects
Description: TTP defined as the time from first dose of study drug until tumor progression as defined by the Revised Recommendations of the International Working Group (IWG) for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia
Time Frame: time from first dose of study drug until tumor progression up to two years after the date of the first documented response.
Population: The study was terminated at Phase I due to Funder's decision
Arm/Group | Phase II:TAK-659 100mg+ Ixazomib MTD
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS) for Phase II Subjects
Description: OS defined as the time from the date of study entry to death
Time Frame: time from the date of study entry up to two years.
Population: This study was terminated at Phase I due to funder's decision
Groups:
- Phase II:TAK-659 100mg+ Ixazomib MTD: Phase II: TAK-659 100 mg (Days 1-15) + Ixazomib at MTD (Days 1, 8, 15)
  TAK-659: Subjects were given 100 mg ofTAK-659 tablets once daily for fifteen days at MTD.
  Ixazomib: Subjects were given Ixazomib capsules once weekly at MTD on days 1, 8,15, respectively at MTD.
  .
Arm/Group | Phase II:TAK-659 100mg+ Ixazomib MTD
Number analyzed (Participants) | 0

6. Secondary Outcome: Frequency of Grade 3 and Higher Adverse Events for Phase II Subjects
Description: Summarize Grade 3 and higher adverse events using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Time Frame: From date of first dose until 30 days after the last treatment up to 1 year.
Population: This study was terminated at Phase I due to funder's decision
Arm/Group | Phase II:TAK-659 100mg+ Ixazomib MTD
Number analyzed (Participants) | 0

7. Secondary Outcome: Mortality Rate at 3 and 6 Months for Phase II Subjects
Description: Number of deaths at 3 and 6 moths are assessed in Phase II subjects.
Time Frame: From start of treatment up to 2 years or until death.
Population: This study was terminated at Phase I due to funder's decision
Arm/Group | Phase II:TAK-659 100mg+ Ixazomib MTD
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the time of consent and for at least 30 days after treatment discontinuation, regardless of whether or not the event(s) were considered related to trial medications. Serious adverse events were reported from the initiation of study drug(s) and for 30 days after administration of the last dose of study drug(s).
Description: Adverse events were collected from the date of first treatment dose until 30 days after the last treatment, assessed for 7 cycles of treatment. Each treatment cycle was of 28 days.
Arm/Group | Phase I, Level 1: TAK-659 100mg + Ixazomid 2.3mg
All-Cause Mortality (participants affected / at risk) | 5/7
Serious Adverse Events (participants affected / at risk) | 5/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Level 1: TAK-659 100mg + Ixazomid 2.3mg (N=7)
DEATH NOS (General disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
HEART FAILURE (Cardiac disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Level 1: TAK-659 100mg + Ixazomid 2.3mg (N=7)
ADULT RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BACTEREMIA (Infections and infestations) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 2 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (5)
BREAST PAIN (Reproductive system and breast disorders) | 1 (3)
CONSTIPATION (Gastrointestinal disorders) | 1 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
EDEMA FACE (General disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FEVER (General disorders) | 2 (3)
FLUSHING (Vascular disorders) | 1 (1)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 1 (1)
GENERALIZED EDEMA (General disorders) | 2 (3)
GGT INCREASED (Investigations) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERPARATHYROIDISM (Endocrine disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 1 (1)
LEUKEMIA SECONDARY TO ONCOLOGY CHEMOTHERAPY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (3)
LIP PAIN (Gastrointestinal disorders) | 1 (1)
LIPASE INCREASED (Investigations) | 2 (3)
LYMPHOCYTE COUNT INCREASED (Investigations) | 3 (3)
MUCOSITIS ORAL (Gastrointestinal disorders) | 3 (4)
NAUSEA (Gastrointestinal disorders) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (3)
ORAL PAIN (Gastrointestinal disorders) | 1 (1)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (2)
PERIORBITAL EDEMA (Eye disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 3 (4)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SERUM AMYLASE INCREASED (Investigations) | 2 (3)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 2 (3)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04079738/Prot_SAP_000.pdf